CLINICAL TRIAL: NCT06631066
Title: Effect of Neoadjuvant Chemoradiation on Pathologic Complete Response Rates in Locally Advanced Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Marwa Mohammmed sayed, assistant lecturer, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RO2109-30909
Record Dates: First submitted 2024-08-13; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Female
Keywords: preoperative radiotherapy; locally advanced breast cancer; pathologic response
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- neoadjuvant chemotherapy arm (No Intervention): The patients in this arm will recieve neoadjuvant chemotherapy (with anti-her2 agents if indicated) according to the national guidelines.
  post systemic treatment imaging will be done to assess the response, followed by surgery as indicated.
  Adjuvant radiotherapy as well as hormonal or target therapy will be prescribed as indicated.
  Radiation therapy will be delivered in hypofractionated course (40.05 Gray over 15 fractions with boost to tumor bed 10 Gray over four fractions) to the breast/ chestwall as well as regional lymphatics.
- Neoadjuvant chemoradiation arm (Experimental): The patients in this arm will recieve neoadjuvant chemotherapy with preoperative radiotherapy concurrently with taxanes. Surgery is done 6-8 weeks as indicated, followed by systemic treatment according to the guidelines.
  Interventions: Radiation: neoadjuvant chemoradiation

INTERVENTIONS:
Radiation: neoadjuvant chemoradiation — Neoadjuvant chemoradiation will be prescribed as: 4 cycles of Adriamycin and Cyclophosphamide followed by radiotherapy concurrently with taxanes/ taxanes and carboplatin. followed by surgery as indicated.
  Arms: Neoadjuvant chemoradiation arm

SUMMARY:
This is a phase II randomized trial comparing pathologic complete response rates in locally advanced patients recieving either neoadjuvant chemotherapy or neoadjuvant chemoradiation.

DETAILED DESCRIPTION:
A prospective randomized phase II trial, that enrolled locally advanced breast cancer patients who were randomized to recieve either neoadjuvant systemic treatment or neoadjuvant systemic treatment concurrently with radiotherapy. Surgery is done for all patients later on as indicated.

The pathological response rates between both groups will be compared, as well as surgical complications and acute radiation toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients.
2. Age: 21 years or older.
3. ECOG performance status (PS) score 0 to 2.
4. Locally advanced tumors (stage IIIA or above) of any subtype.
5. Early breast cancer of the HER2+ or TNBC subtype when:

   1. Node-negative, T2 or T3.
   2. Node-positive, any T stage.

Exclusion Criteria:

1. Patients initially presenting with metastatic breast cancer.
2. Patients unfit to receive planned regimen of treatment that had a poor PS (i.e.: PS 3 and 4).
3. Inflammatory breast cancer (T4d) patients.
4. Patients having contraindications to radiotherapy (e.g.: Pregnancy, history of previous chest wall, breast, or axillary irradiation)
5. History of previous ipsilateral breast surgery.
6. Comorbidities that would affect skin healing or integrity, like uncontrolled diabetes mellitus or active autoimmune collagen or vascular diseases

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 160 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
pathologic complete response rates | 1 week postoperative
  the pathologic response will be measured by the Randomized cancer burden (RCB) scoring system

SECONDARY OUTCOMES:
acute radiation toxicity | during radiation therapy: week 2,3,4. weekly after the end of radiation therapy for 4 weeks
  radiation therapy oncology group (RTOG) acute morbidity score

CONTACTS AND LOCATIONS:
Overall Officials: Medhat El Sebaie, Professor, Study Chair — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ward J, Ho K, Ike C, Wood SH, Thiruchelvam PTR, Khan AA, Leff DR. Pre-operative chemoradiotherapy followed by mastectomy and breast reconstruction-A systematic review of clinical, oncological, reconstructive and aesthetic outcomes. J Plast Reconstr Aesthet Surg. 2024 Sep;96:242-253. doi: 10.1016/j.bjps.2024.07.022. Epub 2024 Jul 15. PMID 39106546
- [Background] O' Halloran N, McVeigh T, Martin J, Keane M, Lowery A, Kerin M. Neoadjuvant chemoradiation and breast reconstruction: the potential for improved outcomes in the treatment of breast cancer. Ir J Med Sci. 2019 Feb;188(1):75-83. doi: 10.1007/s11845-018-1846-6. Epub 2018 Jun 14. PMID 29948462